CLINICAL TRIAL: NCT02183077
Title: Pharmacokinetics and Tolerability of 2 x 15 mg Meloxicam (2 x 0.3 g Topical Gel) Over 7 Days Compared to 7.5 mg Meloxicam Tablet (Single Oral Dose) in Healthy Subjects. A Two-way Cross-over, Randomized, Open Study
Brief Title: Pharmacokinetics and Tolerability of Meloxicam Gel Compared to Meloxicam Tablets in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 107.214
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Meloxicam

ARMS (2):
- Meloxicam gel (Experimental)
  Interventions: Drug: Meloxicam gel
- Meloxicam tablet (Active Comparator)
  Interventions: Drug: Meloxicam tablet

INTERVENTIONS:
Drug: Meloxicam gel
  Arms: Meloxicam gel
Drug: Meloxicam tablet
  Arms: Meloxicam tablet

SUMMARY:
Study to gain information on the percutaneous absorption of meloxicam after administration of a topical gel over 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice and local legislation
* Age >= 18 and <= 50 years
* Broca >= -20% and <= + 20 %

Exclusion Criteria:

* Any findings of the medical examination (including blood pressure, pulse rate and electrocardiogram) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* Hypersensitivity to meloxicam and any of the excipients or non-steroidal antirheumatic agents
* Intake of drugs with a long half-life (>24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the results of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 months prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or >3 pipes/day)
* Inability to refrain from smoking on study days
* Known alcohol abuse
* Known drug abuse
* Blood donation (<= 1 months prior to administration)
* Excessive physical activities (<= 5 days prior to administration)
* History of hemorrhagic diatheses
* History of gastrointestinal ulcer, perforation or bleeding
* History of bronchial asthma
* Any laboratory value outside the normal range of clinical relevance
* History of dermatological diseases
* Skin disease and/or skin lesions at the site of planned application

For female subjects:

* Pregnancy
* Positive pregnancy test
* Breast feeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1998-09; Primary Completion 1998-11 (Actual)

PRIMARY OUTCOMES:
Analysis of plasma concentration-time course after topical dose | up to 264 hours after first topical administration
Determination of the ratio AUCss topical/AUC0-∞ oral | up to 96 hours after oral administration

SECONDARY OUTCOMES:
Maximum measured concentration of the analyte in plasma (Cmax) | up to 96 hours after oral administration
Time from dosing to the maximum concentration of the analyte in plasma (Tmax) | up to 96 hours after oral administration
Total area under the plasma drug concentration time curve (AUC) from time of administration to the time of the last quantifiable drug concentration (AUC0-t) | up to 96 hours after oral administration
Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 96 hours after oral administration
Terminal half-life of the analyte in plasma (t½) | up to 96 hours after oral administration
Apparent terminal elimination rate constant | up to 96 hours after oral administration
Apparent clearance of the analyte in plasma following extravascular administration (CL/F) | up to 96 hours after oral administration
Apparent volume of distribution of the analyte during the terminal phase (Vz/F) | up to 96 hours after oral administration
Mean residence time (MRTtot) | up to 96 hours after oral administration
Excretion of metabolites in urine | 0-24 hours after oral administration
Predose concentration of the analyte in plasma at steady state immediately before administration of the next dose (Cpre,ss) | up to 264 hours after first topical administration
Minimum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmin,ss) | up to 264 hours after first topical administration
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | up to 264 hours after first topical administration
Total area under the plasma drug concentration time curve (AUC) during a steady state interval (AUCss) | up to 264 hours after first topical administration
Terminal half-life of the analyte in plasma (t½) | up to 264 hours after first topical administration
Apparent terminal elimination rate constant | up to 264 hours after first topical administration
Occurence of adverse events | up to 24 days
Assessment of local and systemic tolerability | up to 24 days